CLINICAL TRIAL: NCT05029986
Title: Self-Regulated Airflow Management in Daily Communicative Activities to Prevent Dyspnea During Speech in Older Speakers
Brief Title: Preventing Dyspnea During Speech in Older Speakers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Responsible Party: Principal Investigator, Maude Desjardins, Post-doctoral researcher, University of Delaware
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1767412
Record Dates: First submitted 2021-08-29; First posted 2021-09-01 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Dyspnea
Keywords: dyspnea; speech therapy; communication; aging; breathing; respiratory; intervention; voice
MeSH Terms: conditions — Dyspnea; Communication Disorders; Communication; Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All participants (Experimental): This is a single-arm trial. All participants will receive (1) a control condition (socialization phase, 2 weeks) and (2) an intervention condition (speech breathing intervention, 4 weeks). Group sessions will take place once a week, and participants will be instructed to practice their exercises every day at home during the study duration.
  Interventions: Behavioral: Socialization phase; Behavioral: Speech breathing intervention

INTERVENTIONS:
Behavioral: Socialization phase — Control condition: does not involve speech-related exercises
Behavioral: Speech breathing intervention — Experimental condition: involves speech-related exercises

SUMMARY:
Due to various comorbidities affecting the respiratory system, older speakers are at risk of experiencing breathing discomfort (dyspnea) during high-demand vocal activities such as singing, loud speaking, and speaking while exercising. Dyspnea during speech can promote avoidance of certain situations involving voice production, thus leading to vocal deconditioning and decreased quality of life. The goal of this pilot study is to test the feasibility and acceptability of a 4-week remote group intervention targeting phonatory dyspnea, and to gather preliminary efficacy data.

Participants will receive an intervention including a 2-week socialization phase (control condition) and a 4-week speech breathing intervention phase (experimental condition). Both phases will be delivered remotely and in a group setting (10 participants per group).

ELIGIBILITY:
Inclusion Criteria:

* sign the informed consent form
* report dyspnea in at least one of the items of the University of Cincinnati Dyspnea Questionnaire referring to speech
* be available during the dates of the scheduled group interventions
* be aged 50 years or older

Exclusion Criteria:

* do not have access to a computer and internet connection
* present with a known voice pathology (other than age-related vocal fold atrophy) and/or are receiving speech therapy at the time of the study
* have a known neurodegenerative disease affecting speech/voice
* are a current smoker
* are receiving pulmonary rehabilitation at the time of the study or are starting a new medication regimen for a respiratory disease at the time of study onset;
* have a hearing loss that is not adequately managed, as judged by the Principal Investigator (PI)
* have professional vocal training [amateur choir singers will not be excluded]
* cannot provide informed consent or easily follow instructions
* have any other condition that precludes them from participating in the behavioral interventions, as judged by the PI.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2022-03-10 (Actual); Study Completion 2022-03-10 (Actual)

PRIMARY OUTCOMES:
Change in reported dyspnea | Assessed at baseline, after the 2-week control condition, and after the 4-week experimental condition.
  Participant self-ratings of dyspnea on the University of Cincinnati Dyspnea Questionnaire. This questionnaire contains 30 items scored on a Likert scale ranging from 1 (not at all short of breath) to 5 (always short of breath or cannot do). A higher scores indicates greater shortness of breath and therefore greater handicap.
Change in reported voice handicap | Assessed at baseline, after the 2-week control condition, and after the 4-week experimental condition.
  Participant self-ratings of voice handicap on the Voice Handicap Index-10. The Voice Handicap Index-10 is an ordinal scale that measures the degree of handicap a person experiences because of their voice disorder. Each item is scored on a Likert scale ranging from 0 to 4. The minimum score is 0 and the maximal score 40. A higher score indicates a greater perceived voice handicap.

SECONDARY OUTCOMES:
Change in reported self-efficacy | Assessed at baseline, after the 2-week control condition, and after the 4-week experimental condition.
  Participant self-ratings of self-efficacy for managing their symptoms, using the Patient-Reported Outcomes Measurement Information System (PROMIS) Self-Efficacy Questionnaire - Managing Symptoms. This questionnaire contains 28 items, each scored on a Likert scale ranging from 1 (I am not at all confident) to 5 (I am very confident). A higher score indicates a greater self-efficacy.
Acceptability of the intervention | Assessed after the 4-week experimental condition, at the end of the study period.
  Participants' perceived acceptability of the intervention using the Acceptability of Intervention Measure. This questionnaire contains 5 items scored on a Likert scale ranging from 1 (completely disagree) to 5 (completely agree). A higher score indicates a greater acceptability.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Delaware, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: No